CLINICAL TRIAL: NCT04053855
Title: Evaluation of Urinary Exosomes Presence From Clear Cell Renal Cell Carcinoma
Acronym: PEP-C
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 19CH048; 2019-A01408-49 (Other: ANSM)
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: Clear cell renal cell carcinoma; Urinary exosomes; Detection; Electron microscopy technique; Flow cytometry; RT-qPCR
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urinary sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Renal mass patients: Patients with renal mass requiring surgery (partial or total nephrectomy) will be included.
  They will have an urinary sample.
  Interventions: Biological: Urinary sample
- Control patients: Control patients (without renal mass) will be included. They will have an urinary sample.
  Interventions: Biological: Urinary sample

INTERVENTIONS:
Biological: Urinary sample — Urinary sample (100 ml) will be collected in the urology department to analysis urinary exosomes.

SUMMARY:
Clear cell renal cell carcinoma is diagnosed by imaging, sometimes associated with biopsy. This diagnosis is expensive, invasive and sometimes late. The development of a simple biological test for diagnosis is essential. Exosomes are 30 to 150 nm membrane vesicles secreted into the extracellular space by various living cells. These exosomes can be isolated from biological fluids, including urine. The recent study of urinary exosomes is a promising topic for analyzing tumor markers in urine. The investigator's goal is to develop a reliable technique for detecting tumor exosomes in urine in patients with clear cell renal cell carcinoma. The analysis of urinary exosomes could provide a new liquid biopsy tool for the early diagnosis of clear cell renal cell carcinoma.

DETAILED DESCRIPTION:
The primary objective is to detect urinary exosomes, by electron microscopy technique, from clear cell renal cell carcinoma due to exosome markers (CD9) and clear cell kidney cancer (CA9).

ELIGIBILITY:
Inclusion Criteria:

Patients:

* All patients with renal mass requiring surgery (partial or total nephrectomy)
* Social security affiliation
* Signed informed consent

Control :

* Unscheduled nephrectomy
* Social security affiliation
* Signed informed consent

Exclusion Criteria:

* Insufficient volume of urine sample (< 100 ml)
* Patients with a urinary catheter
* Patients under court-ordered guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients and 40 control will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients (with clear cell kidney cancer) with CD9+ and CA9+ exosomes by electron microscopy technique | At inclusion
  Measured by analysis in electron microscopy technique of urinary sample.

SECONDARY OUTCOMES:
Percentage of CD9+ /CA9+ exosomes by electron microscopy technique (%) for patients with clear cell kidney cancer | At inclusion
  Measured by analysis in electron microscopy technique of urinary sample.
Percentage of CD9+ /CA9+ exosomes by electron microscopy technique (%) for control patients | At inclusion
  Measured by analysis in electron microscopy technique of urinary sample.
Percentage of CD9+ /CA9+ exosomes by flow cytometry (%) for patients with clear cell kidney cancer | At inclusion
  Measured by analysis in flow cytometry of urinary sample.
Percentage of CD9+ /CA9+ exosomes by flow cytometry (%) for control patients | At inclusion
  Measured by analysis in flow cytometry of urinary sample.
Percentage of CD9+ /CA9+ exosomes by Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) (%) for control patients | At inclusion
  Measured by analysis in Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) of urinary sample.
Percentage of CD9+ /CA9+ exosomes by Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) (%) for patients with clear cell kidney cancer | At inclusion
  Measured by analysis in Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) of urinary sample.
Percentage of CD9+/CD63+/CD81+/CA9+ exosomes by electron microscopy technique (%) for patients with clear cell kidney cancer | At inclusion
  Measured by analysis in electron microscopy technique of urinary sample.
Percentage of CD9+/CD63+/CD81+/CA9+ exosomes by electron microscopy technique (%) for control patients | At inclusion
  Measured by analysis in electron microscopy technique of urinary sample.
Percentage of CD9+/CD63+/CD81+/CA9+ exosomes by flow cytometry (%) for patients with clear cell kidney cancer | At inclusion
  Measured by analysis in flow cytometry of urinary sample.
Percentage of CD9+/CD63+/CD81+/CA9+ exosomes by flow cytometry (%) for control patients | At inclusion
  Measured by analysis in flow cytometry of urinary sample.
Percentage of CD9+/CD63+/CD81+/CA9+ exosomes by Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) (%) for patients with clear cell kidney cancer | Years: 2
  Measured by analysis in Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) of urinary sample.
Percentage of CD9+/CD63+/CD81+/CA9+ exosomes by Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) (%) for control patients | Years: 2
  Measured by analysis in Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) of urinary sample.
Percentage of CD9+/VGEFR2+ exosomes by electron microscopy technique (%) for patients with clear cell kidney cancer | At inclusion
  Measured by analysis in electron microscopy technique of urinary sample.
Percentage of CD9+/VGEFR2+ exosomes by electron microscopy technique (%) for control patients | At inclusion
  Measured by analysis in electron microscopy technique of urinary sample.
Percentage of CD9+/VGEFR2+ exosomes by flow cytometry (%) for patients with clear cell kidney cancer | At inclusion
  Measured by analysis in flow cytometry of urinary sample.
Percentage of CD9+/VGEFR2+ exosomes by flow cytometry (%) for control patients | At inclusion
  Measured by analysis in flow cytometry of urinary sample.
Percentage of CD9+/VGEFR2+ exosomes by Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) (%) for patients with clear cell kidney cancer | At inclusion
  Measured by analysis in Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) of urinary sample.
Percentage of CD9+/VGEFR2+ exosomes by Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) (%) for control patients | At inclusion
  Measured by analysis in Reverse Transcription quantitative Polymerase Chain Reaction (RT-qPCR) of urinary sample.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MOTTET, MD PhD, Principal Investigator — CHU SAINT-ETIENNE; Nora MALLOUK, PhD, Study Chair — UNIVERSITY SAINT-ETIENNE; Guorong LI, PhD, Study Chair — CHU DE SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li G, Mallouk N, Flandrin P, Garcin A, Lambert C, Berremila SA, Habchi H, Mottet N. Presence of Urinary Exosomes for Liquid Biopsy of Clear Cell Renal Cell Carcinoma: Protocol for a Pilot Feasibility Study. JMIR Res Protoc. 2021 Jul 20;10(7):e24423. doi: 10.2196/24423. PMID 34283029